CLINICAL TRIAL: NCT06685848
Title: Multi-Center, Randomized, Controlled Cross-Over Study to Evaluate Safety and Effectiveness of Hypoxic RBCs Processed With the Hemanext ONE System vs Conventional RBCs in Patients With Transfusion-Dependent Haematological Malignancies
Brief Title: Comparison of Hemanext ONE® System and Conventional Red Blood Cell Transfusion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hemanext (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PRO-CLIN-0015
Record Dates: First submitted 2024-11-05; First posted 2024-11-13 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Hematologic Neoplasms
Keywords: Transfusion; Red Blood Cells; Hypoxic
MeSH Terms: conditions — Hematologic Neoplasms; Hypoxia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- A - Hemanext ONE system (Experimental): Hypoxic RBCs
  Interventions: Device: Hemanext ONE system
- B - Conventional RBCs (Active Comparator): Conventional RBCs
  Interventions: Device: Conventional RBCs

INTERVENTIONS:
Device: Hemanext ONE system — Hypoxic red blood cells
  Arms: A - Hemanext ONE system
Device: Conventional RBCs — Conventional manufactured Red blood cells
  Arms: B - Conventional RBCs

SUMMARY:
The overall objective of this study is to collect preliminary effectiveness and safety data on the transfusion of hypoxic RBCs, manufactured with the Hemanext ONE device, in patients with hematological malignancies. The Hemanext ONE device received CE mark in April 2021.

DETAILED DESCRIPTION:
The primary objective is to evaluate whether the total number of hypoxically stored red blood cell (RBCs) units per unit of time transfused in patients with haematologic malignancies, requiring chronic blood transfusion therapy, is non-inferior to the total number of units of conventionally stored RBCs per unit of time transfused.

Secondary objectives include the following:

1. Analysis of volume of blood transfused
2. Analysis of number of transfusion events throughout the study period
3. Key laboratory assessments (hemoglobin and hematocrit) and average hemoglobin increment after transfusions of hypoxically stored RBCs compared to that with conventionally stored RBCs
4. Evaluation of Quality of Life (QoL)
5. Change in serum ferritin
6. Safety assessment

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 or older
* Patients with a documented diagnosis of a haematological malignancy requiring chronic transfusions.
* If MDS patient, Have low risk or intermediate risk MDS per either IPSS-R (https://www.mds-foundation.org/ipss-r-calculator/) or IPSS-M (IPSS-M Risk Calculator (mds-risk-model.com))
* If MDS patient, a bone marrow aspirate completed within the 6 months prior to study enrolment, and which did not show progression to higher risk MDS
* Have RBC transfusion dependence (at least 2 RBC units /8 weeks during the last 16 weeks)
* Baseline RBC transfusion threshold of 9 g/dL
* ECOG (Eastern Cooperative Oncology Group) performance status < 3
* Have signed the informed consent form and are willing to comply with the study visits and procedures
* If on Iron Chelation Therapy, have been on a stable dose for ≥3 months prior to screening

Exclusion Criteria:

* Have a life expectancy of less than 1 year
* Have palpable splenomegaly (more than 3 cm below the mid clavicular line)
* Have other associated causes of anemia (including auto-immune hemolysis or active hemorrhage, or progression to acute leukemia)
* If prescribed erythropoiesis affecting disease modifying agents (e.g. G-CSF, erythropoietin), have not been on a stable dose for 90 days
* Is currently taking Luspatercept or other investigational erythropoiesis affecting disease modifying agent
* Have severe renal insufficiency with creatinine clearance (MDRD or CKD EPI) below 30ml/min
* Have lung disease with hypoxia or oxygen-dependent
* Have severe coronary artery disease (including unstable angina or recent myocardial infraction) or severe heart failure (left ventricular ejection fraction less than 30%)
* Have a history of cancer active in the previous 3 years, except local cervix cancer, or basal cell cutaneous carcinoma
* Have a history of allo-immunization other than rhesus Kell that cannot be managed by the local blood bank
* Are a female of child-bearing potential that is pregnant, planning to become pregnant in the next 14 months or breastfeeding
* Are a patient under guardianship or curatorship
* Are currently participating in another interventional study evaluating an erythropoiesis affecting disease modifying agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-11-29 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Number of RBCs units per unit of time | Through study completion, an average of 15 months
  The difference in the total number of hypoxic RBCs units per unit of time transfused to MDS patients during the study period compared to the total number of conventional RBCs units per unit of time transfused.

SECONDARY OUTCOMES:
Volume of blood transfused | Through study completion, an average of 15 months
  The mean volume of blood per patient transfused with Hemanext ONE and with standard RBC units will be analyzed and compared
Number of transfusion events | Through study completion, an average of 15 months
  Mean number of transfusion events throughout the study period
Mean change in key laboratory assessments (hemoglobin) | Up to 15-60 minutes post transfusion, up to day 7, up to pre-transfusion of first washout visit (at 6 months), up to transfusion on the final transfusion visit (at 15 months)
  Mean change in key laboratory assessments (hemoglobin) and average hemoglobin increment after transfusions of hypoxically stored RBCs compared to that with conventionally stored RBCs.
Mean change in key laboratory assessments (hematocrit) | Up to 15-60 minutes post transfusion, up to day 7, up to pre-transfusion of first washout visit (at 6 months), up to transfusion on the final transfusion visit (at 15 months)
  Mean change in key laboratory assessments (hematocrit) after transfusions of hypoxically stored RBCs compared to that with conventionally stored RBCs.
Mean change in QoL | At the end of first transfusion cycle at 6 months and at study exit (at 15 months)
  Mean change in QoL as assessed by the EORTC QLQ-C30 (EORTC Quality of Life Questionnaire).
  Scores from 1-4 (where 1 indicates a better outcome and 4 indicates a worse outcome):
  1. Not at all
  2. A little
  3. Quite a bit
  4. Very Much
  Additionally, a rating from 1-7, where 1 is "Very poor" and 7 is "Excellent"
Mean change in serum ferritin | At the end of first transfusion cycle at 6 months and at study exit (at 15 months)
  Mean change from baseline in serum ferritin (assessment during baselines 1 and 2 (first pre-transfusion visit of each arm) to pre-transfusion of first washout visit and pre-transfusion of the final visit).
Safety assessment in terms of frequency of adverse event reactions and device deficiencies. | Through study completion, an average of 15 months
  Safety assessment in terms of frequency of adverse event reactions and device deficiencies.

CONTACTS AND LOCATIONS:
Overall Officials: Håkon Reikvam, PhD, MD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No